CLINICAL TRIAL: NCT06737913
Title: Hepatic Arterial Infusion or Intravenous Infusion of Adebrelimab, Combined with Bevacizumab and Hepatic Arterial Infusion of FOLFOX Chemotherapy for Advanced Hepatocellular Carcinoma: a Multicenter, Open Label, Randomized Phase II Trial
Brief Title: HAI or IV of Adebrelimab, Combined with Bevacizumab and HAI of FOLFOX for Advanced Unresectable Hepatocellular Carcinoma
Acronym: HAIBrave-001
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Henan Provincial People's Hospital (Other); First Affiliated Hospital of Fujian Medical University (Other); Shanghai Zhongshan Hospital (Other); Cancer Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Weijun Fan, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2024-588-01; ChiCTR2400092928 (Other: Chinese Clinical Trial Register)
Record Dates: First submitted 2024-12-11; First posted 2024-12-17 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Advanced Hepatocellular Carcinoma (HCC)
Keywords: Hepatic arterial infusion (HAI); hepatic arterial infusion of FOLFOX chemotherapy; advanced unresectable hepatocellular carcinoma (HCC); Adebrelimab (ADE); Bevacizumab (Bev.); intravenous infusion (IV)
MeSH Terms: interventions — Bevacizumab; Infusions, Intravenous; Folfox protocol

STUDY DESIGN:
Intervention Model Description: A total of 78 patients (anticipated) will be randomized (1:1) to two arms to receive Hepatic arterial infusion (HAI) of Adebrelimab (ADE) (1200mg, IA, Q3W) and intravenous infusion (IV) of Bevacizumab (Bev.) (15mg/kg, IV, Q3W) plus HAIC with FOLFOX regimen (oxaliplatin 85 mg/m2, leucovorin 400 mg/m2, 5-fluorouracil bolus 400 mg/m2 on day 1, and 5-fluorouracil infusion 2500 mg/m2 for 46 hours via hepatic artery Q4W) or intravenous infusion (IV) of Adebrelimab (ADE) (1200mg, IV, Q3W) and intravenous infusion (IV) of Bevacizumab (Bev.) (15mg/kg, IV, Q3W) plus HAIC with FOLFOX regimen (oxaliplatin 85 mg/m2, leucovorin 400 mg/m2, 5-fluorouracil bolus 400 mg/m2 on day 1, and 5-fluorouracil infusion 2500 mg/m2 for 46 hours via hepatic artery, Q3W). The Two arms continue the triple combination treatment up to 6 cycles and then received receive intravenous combination therapy of adebrelimab and bevacizumab for maintainance until disease progression or intolerable toxicity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HAIBrave-001 Arm 1 (Experimental): Arm 1 to receive Hepatic arterial infusion (HAI) of Adebrelimab (ADE) + intravenous infusion (IV) of Bevacizumab (Bev.) + Hepatic artery infusion chemotherapy (HAIC) with FOLFOX regimen
  Interventions: Procedure: HAI Adebrelimab; Drug: intravenous infusion (IV) of Bevacizumab (Bev.); Procedure: HAIC with FOLFOX regimen; Drug: Adebrelimab and bevacizumab maintainance treatment
- HAIBrave-001 Arm 2 (Experimental): Intravenous infusion (IV) of Adebrelimab (ADE) + intravenous infusion (IV) of Bevacizumab (Bev.)+ HAIC with FOLFOX regimen
  Interventions: Drug: intravenous infusion (IV) of Adebrelimab (ADE); Drug: intravenous infusion (IV) of Bevacizumab (Bev.); Procedure: HAIC with FOLFOX regimen; Drug: Adebrelimab and bevacizumab maintainance treatment

INTERVENTIONS:
Procedure: HAI Adebrelimab — Hepatic arterial infusion (HAI) of Adebrelimab (ADE) (1200mg, IA, Q3W)
  Other Names: HAI FOLFOX; IV Bevacizumab; IV Adebrelimab
  Arms: HAIBrave-001 Arm 1
Drug: intravenous infusion (IV) of Adebrelimab (ADE) — intravenous infusion (IV) of Adebrelimab (ADE) (1200mg, IV, Q3W)
  Arms: HAIBrave-001 Arm 2
Drug: intravenous infusion (IV) of Bevacizumab (Bev.) — intravenous infusion (IV) of Bevacizumab (Bev.) (15mg/kg, IV, Q3W)
Procedure: HAIC with FOLFOX regimen — HAIC with FOLFOX regimen (oxaliplatin 85 mg/m2, leucovorin 400 mg/m2, 5-fluorouracil bolus 400 mg/m2 on day 1, and 5-fluorouracil infusion 2500 mg/m2 for 46 hours via hepatic artery Q4W)
Drug: Adebrelimab and bevacizumab maintainance treatment — The two arms continue the triple combination treatment up to 6 cycles and then received receive intravenous combination therapy of adebrelimab and bevacizumab for maintainance until disease progression or intolerable toxicity

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Adabrelimab (arterial or intravenous administration) combined with hepatic artery FOLFOX infusion chemotherapy and Bevacizumab as the first-line treatment of advanced stage hepatocellular carcinoma. Patients will be randomized 1:1 etither to receive hepatic arterial infusion(HAI) Adabrelimab group or IV Adabrelimab group, and both groups will receive HAI FOLFOX chemotherapy and IV Bevacizumab.

DETAILED DESCRIPTION:
The combination of anti-PD-L1 antibody and bevacizumab has been approved as the first-line treatment for advanced hepatocellular carcinoma (HCC). However, the overall response rate is still unsatisfactory and the prognosis of patients remains poor. Our previous retrospective analysis showed triple combination of hepatic arterial infusion chemotherapy (HAIC) of FOLFOX regimen plus adebrelimab (anti-PD-L1 antibody) and bevacizumab had a high response rate for advanced stage HCC patients. More, as the PD-L1 on intrahepatic tumors is the main target of anti-PD-L1 therapy, hepatic arterial infusion of anti-PD-L1 antibody may contribute to a synergistic effect. Herein, we aimed to evaluate the efficacy and safety of Adabrelimab (arterial or intravenous administration) combined with hepatic artery FOLFOX infusion chemotherapy and Bevacizumab as the first-line treatment of advanced stage hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the study and sign the informed consent form; 2, Aged ≥18 years (calculated as of the date of signing the informed consent form); 3 .Diagnosed with hepatocellular carcinoma (HCC) by clinical or pathological means; 4. Barcelona Clinic Liver Cancer (BCLC) stage C, with vascular/bile duct invasion or distant metastasis (excluding cases with Vp4-type tumor thrombus); 5. No prior systemic therapy for HCC; or progression or residual lesions following prior local therapy for HCC (including but not limited to surgery, ablation, radiotherapy, or transarterial chemoembolization [TACE]), with an interval of at least one month between the last local treatment and enrollment; 6. ECOG Performance Status (PS) score of 0-1 and Child-Pugh grade A or grade B with a score of 7; 7. No history of autoimmune disease; 8. An expected survival time of ≥3 months; 9. At least one measurable lesion (per RECIST v1.1 criteria, the longest diameter of the measurable lesion on spiral CT scan must be ≥10 mm or the short axis of enlarged lymph nodes must be ≥15 mm; lesions previously treated locally can be considered target lesions if progression is confirmed per RECIST v1.1 criteria); 10. Sufficient hematologic, hepatic, and renal function, with laboratory tests within the following parameters performed within one week prior to enrollment:

* Neutrophil count ≥1.5×10^9/L;

  * Platelet count ≥75×10^9/L; ③ Hemoglobin ≥90 g/L;

    * Serum ALT and AST ≤5×upper limit of normal (ULN);

      * Serum creatinine ≤1.5×ULN;

        * International Normalized Ratio (INR) <2.3, or prothrombin time ≤ULN+6 seconds;

          * Albumin ≥30 g/L; ⑧ Total bilirubin ≤3×ULN. 11.Women of childbearing potential must have a negative serum or urine pregnancy test within seven days prior to study enrollment, must not be breastfeeding, and must agree to use contraceptive measures during the study and for six months after its conclusion; men must agree to use contraceptive measures during the study and for six months after its conclusion.

Exclusion Criteria:

1. Patients with a severe allergy to iodine contrast agents who are unable to undergo hepatic arterial infusion chemotherapy (HAIC);
2. Use of immunosuppressants or systemic corticosteroids for immunosuppressive purposes within one month prior to randomization;
3. Active infections that cannot be effectively controlled;
4. Severe gastroesophageal varices; untreated or incompletely treated gastroesophageal varices (with bleeding or high risk of bleeding);
5. Presence of brain metastases or bone metastases requiring urgent surgical or radiotherapy intervention;
6. Pregnant or suspected to be pregnant, or currently breastfeeding;
7. Current use or recent use (within 10 days before the initiation of the study treatment) of aspirin (>325 mg/day, maximum antiplatelet dose) or dipyridamole, ticlopidine, clopidogrel, and cilostazol;
8. Thrombotic or embolic events, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, or cerebral infarction) or pulmonary embolism, occurring within six months prior to the initiation of the study treatment;
9. Congenital or acquired immunodeficiency;
10. History of other malignant tumors;
11. Any of the following conditions within 12 months prior to the initiation of the study: myocardial infarction, severe/unstable angina, or congestive heart failure;
12. Renal insufficiency requiring dialysis;
13. History of organ transplantation;
14. Severe acute or chronic physical or mental illnesses or laboratory abnormalities that may increase study risks or interfere with result interpretation, rendering the patient unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 6 weeks
  Defined as the proportion of enrolled patients in each group who achieve either a complete response (CR) or partial response (PR) as the best response during the study, based on RECIST v1.1 criteria. Radiology imaging evaluations will be conducted every 6 weeks (or after every two treatment cycles) to assess treatment efficacy.

SECONDARY OUTCOMES:
Progression-free survival (PRS) | 36 months
  The time from the start of treatment to the first occurrence of disease progression based on RECIST 1.1 criteria or death.
Overall survival(OS) | 36 months
  Overall Survival (OS): Patient survival status will be regularly monitored through on-site visits or telephone follow-ups after the end of study treatment until death. If a participant dies during the study, the actual time of death will be recorded.
Time to progression | 36 months
  Time from the date of initial treatment to disease progression based on RECIST 1.1 criteria.
Disease control rate | 36 months
  The proportion of patients with best response of complete remission, partial remission or stable disease based on RECIST 1.1 criteria.
Duration of response | 36 months
  Refer to the time from the first documentation of complete remission or partial remission to the time of imaging-based disease progression based on RECIST 1.1 criteria.
Best overall response | 36 months
  Refer to the best overall response between the date of enrollment to the date of disease progression or the initiation date of other sequential treatments.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No